CLINICAL TRIAL: NCT07264036
Title: Injectable Augmentation Outcomes in Post-Radiation Head and Neck Cancer Patients With Velopharyngeal Dysfunction
Brief Title: Velopharyngeal Dysfunction in Head & Neck Cancer Patients, Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanessa Torrecillas (Other)
Responsible Party: Sponsor-Investigator, Vanessa Torrecillas, Assistant Professor of Otolaryngology - Head & Neck Surgery, University of Virginia
Organization: University of Virginia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PJ05069
Record Dates: First submitted 2025-11-17; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Velopharyngeal Insufficiency; Head and Neck Cancer; Survivorship; Dysphagia; Speech Disorder
Keywords: velopharyngeal dysfunction; hypernasal speech; pharyngeal wall augmentation; nasometry; head and neck cancer; survivorship
MeSH Terms: conditions — Velopharyngeal Insufficiency; Head and Neck Neoplasms; Deglutition Disorders; Speech Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic with Possible Injection Augmentation (Experimental): All participants will undergo a standardized, multidisciplinary evaluation including physical examination, flexible nasolaryngoscopy, acoustic speech analysis, nasometry, clinical swallowing assessment, and fiberoptic endoscopic evaluation of swallowing (FEES). A subset of participants with confirmed velopharyngeal dysfunction (VPD) who meet clinical criteria may elect to receive a pharyngeal wall augmentation injection as part of standard-of-care treatment. All participants, regardless of whether they receive the injection, will have pre-assessment data collected to evaluate speech intelligibility, nasalance, swallowing function, and patient-reported outcomes. The patients who undergo the pharyngeal augmentation injection will also have post-assessment data collected. No formal comparison between participants who do and do not receive the injection will be performed; all data will be analyzed individually.
  Interventions: Procedure: Pharyngeal Wall Augmentation Injection

INTERVENTIONS:
Procedure: Pharyngeal Wall Augmentation Injection — Participants with confirmed velopharyngeal dysfunction (VPD) who meet clinical criteria may elect to receive a pharyngeal wall augmentation injection. The procedure involves the submucosal injection of a biocompatible material into the posterior pharyngeal wall to improve velopharyngeal closure during speech and swallowing. Injection volume and technique will be determined by the treating clinician based on individual anatomy and functional assessment. All participants will undergo standardized assessments of speech intelligibility, nasalance, swallowing function, and patient-reported outcomes before and after the procedure.
  Timing:
  The procedure will occur once at the clinically indicated visit. Post-procedure assessments will be conducted at standardized follow-up intervals to evaluate functional outcomes

SUMMARY:
Some head and neck cancer survivors develop velopharyngeal dysfunction (VPD), a problem with closure between the soft palate and throat that can cause nasal-sounding speech, food or liquid leaking into the nose, difficulty swallowing, and reduced quality of life. This study aims to better understand VPD in this population and to evaluate whether pharyngeal wall augmentation (plumping up the back wall of the throat) can improve speech and swallowing.

Participants will undergo a multidisciplinary assessment including physical examination, flexible nasolaryngoscopy, speech recording and acoustic analysis, nasometry, clinical swallowing evaluation, and fiberoptic endoscopic evaluation of swallowing (FEES).

Aim 1: Determine the prevalence, severity, and functional impact of VPD in head and neck cancer survivors.

Aim 2: Assess the feasibility and usefulness of advanced diagnostic tools for VPD.

The investigators hypothesize that high nasalance scores (>1 SD above normal) will accurately predict VPD with at least 75% positive predictive value and will correlate with worse communication-related quality of life (CPIB).

The investigators also hypothesize that participants with VPD will have more pharyngeal residue or nasal regurgitation on FEES, and that these findings will be associated with lower swallowing-related quality of life (SWAL-QOL).

Aim 3: Evaluate the effectiveness of pharyngeal wall augmentation injections for improving speech intelligibility and swallowing function.

The investigators expect that this treatment will lead to measurable changes in both objective assessments and patient-reported outcomes. The results will help improve diagnosis and management of VPD in head and neck cancer survivors.

DETAILED DESCRIPTION:
Velopharyngeal dysfunction (VPD) is a disorder in which the soft palate and posterior pharyngeal wall do not close adequately during speech and swallowing. Head and neck cancer (HNC) survivors may develop VPD as a result of neuromuscular impairment from surgical resection and/or radiation therapy. Consequences include hypernasal speech from nasal air escape, nasopharyngeal residue during swallowing, nasal regurgitation, and reductions in speech and swallowing-related quality of life. Despite its clinical relevance, VPD in HNC survivors is under-recognized, and evidence regarding optimal diagnostic methods and effective interventions remains limited. This study aims to characterize VPD in this population, evaluate the diagnostic utility of advanced assessment tools, and assess the therapeutic effect of pharyngeal wall augmentation.

Overview This is a prospective study using a multidisciplinary, multimodal assessment protocol to evaluate speech and swallowing function in HNC survivors with suspected or confirmed VPD. Participants will undergo standardized clinical, instrumental, and patient-reported outcome assessments. A subset of participants with confirmed VPD will receive pharyngeal wall augmentation as part of standard clinical care, allowing for pre- and post-intervention comparison.

Aim 1: Characterization of VPD in HNC Survivors

Describe the prevalence, severity, and functional impact of VPD in this population. Participants will complete a comprehensive evaluation including:

Oropharyngeal physical examination to identify structural or neuromuscular contributors to impaired velopharyngeal closure.

Flexible nasolaryngoscopy to assess closure patterns during speech and swallowing tasks.

Acoustic speech analysis and objective measures of speech intelligibility.

Nasometry to quantify nasalance and the degree of hypernasality.

Clinical swallowing evaluation, documenting perceptual indicators of safety and efficiency.

Fiberoptic Endoscopic Evaluation of Swallowing (FEES) to visualize bolus flow, pharyngeal residue, and nasal regurgitation.

Patient-reported outcomes will include the Speech Handicap Index (SHI) and the Swallowing Quality of Life Questionnaire (SWAL-QOL). These measures will characterize functional limitations associated with VPD.

Aim 2: Feasibility and Utility of Advanced Diagnostic Tools Aim 2a: Nasometry as a Diagnostic Indicator This component evaluates whether nasalance scores can reliably identify VPD. The primary hypothesis is that nasalance values >1 standard deviation above normative means will demonstrate a positive predictive value ≥75% when compared with endoscopic confirmation. Correlations will be assessed between nasalance and SHI scores to determine whether acoustic measures reflect patient-perceived communication limitations.

Aim 2b: FEES Indicators of VPD and Functional Correlates

This component assesses whether swallowing abnormalities on FEES are associated with VPD. Participants with confirmed VPD are expected to exhibit:

increased pharyngeal residue, and/or nasal regurgitation during bolus presentation.

These findings will be correlated with SWAL-QOL scores to determine whether FEES characteristics reflect functional swallowing impairment. Results may support FEES as a useful adjunctive tool in evaluating the impact of VPD on swallowing physiology.

Aim 3: Efficacy of Pharyngeal Wall Augmentation Participants with confirmed VPD who are clinically indicated for treatment will undergo pharyngeal wall augmentation using standard-of-care techniques. Injection material and volume will be determined by treating clinicians. The intervention is intended to reduce the velopharyngeal gap and improve closure during speech and swallowing.

Outcome Measures

Pre- and post-intervention comparisons will include:

Nasalance scores Acoustic speech parameters and overall intelligibility Perceptual ratings of speech resonance FEES findings (pharyngeal residue, nasal regurgitation) Patient-reported outcomes (SHI, SWAL-QOL) Participant-reported impressions of change

The primary hypothesis is that pharyngeal wall augmentation will result in measurable improvement in both objective assessments and patient-reported function.

Significance

This study will provide:

A comprehensive description of VPD in HNC survivors. Evidence on the diagnostic value of nasometry and FEES for identifying clinically meaningful VPD.

Prospective data on the functional impact of pharyngeal wall augmentation. Findings will inform best practices for the diagnosis and management of VPD in HNC survivors and support the development of multidisciplinary clinical pathways for improving communication and swallowing outcomes.

ELIGIBILITY:
Inclusion Criteria:

English-speaking adults (≥18 years) History of head and neck cancer treated with surgical resection, chemoradiation, or both Presence of perceptual hypernasality on clinical assessment

Exclusion Criteria:

Pre-existing or suspected non-cancer-related causes of velopharyngeal dysfunction Contraindications to pharyngeal wall augmentation Requirement for more intensive active cancer surveillance Planned future surgical or medical treatments to the pharynx that would interfere with participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Nasometry and FEES for Characterizing Velopharyngeal Dysfunction | Baseline Assessment
  Feasibility will be reported as the percentage of enrolled participants with complete, usable nasometry and FEES data at baseline. Data quality will be defined by the proportion of recordings meeting predefined technical standards for interpretation. Additional exploratory analyses will examine correlations between nasometry and FEES findings and clinical reference standards (perceptual speech ratings, SHI and SWAL-QOL scores), but correlation statistics will not be used as outcome units for feasibility reporting.

SECONDARY OUTCOMES:
Accuracy of Nasometry for Identifying VPD | Baseline
  Proportion of participants with elevated nasalance scores (>1 SD above normative mean) who also demonstrate VPD on flexible nasopharyngoscopy as determined by skilled rater.
Nasometry Characterization of Velopharyngeal Dysfunction | Baseline, 6 weeks post injection
  Nasalance will be quantified using nasometry (percent resonance score). Higher values indicate greater hypernasality.
Modified FEES Observation of Pharyngeal Residue and Nasal Regurgitation | Baseline, 6 weeks post injection
  Proportion of participants demonstrating residue or nasal regurgitation on modified FEES exam.
Patient-Reported Communication Function | Baseline, 6 weeks post injection, 6 months post injection
  Change in total Speech Handicap Index (SHI) score
Change in Patient Reported Swallowing-Related Quality of Life | Baseline, 6 months post injection, 6 months post injection
  SWAL-QOL total score

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Torrecillas, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Study results will be published in peer-reviewed journals. Individual participant-level data will not be made publicly available. Only aggregate data and summary findings will be shared.

REFERENCES:
- [Background] Youssof S, Romero-Clark C, Warner T, Plowman E. Dysphagia-related quality of life in oculopharyngeal muscular dystrophy: Psychometric properties of the SWAL-QOL instrument. Muscle Nerve. 2017 Jul;56(1):28-35. doi: 10.1002/mus.25441. Epub 2017 Feb 12. PMID 27759888
- [Background] Starmer HM, Tippett DC, Webster KT. Effects of laryngeal cancer on voice and swallowing. Otolaryngol Clin North Am. 2008 Aug;41(4):793-818, vii. doi: 10.1016/j.otc.2008.01.018. PMID 18570960
- [Background] Neubauer PD, Rademaker AW, Leder SB. The Yale Pharyngeal Residue Severity Rating Scale: An Anatomically Defined and Image-Based Tool. Dysphagia. 2015 Oct;30(5):521-8. doi: 10.1007/s00455-015-9631-4. Epub 2015 Jun 7. PMID 26050238
- [Background] Kummer, A. W. (2014). Evaluation and treatment of resonance disorders. Language, Speech, and Hearing Services in Schools, 45(3), 183-195. https://doi.org/10.1044/2014_LSHSS-14-0036
- [Background] Karnell, M. P., Christensen, A. J., & Rosenthal, E. L. (2007). Quality of life outcomes in head and neck cancer patients post-treatment. Otolaryngology-Head and Neck Surgery, 136(5), 698-703. https://doi.org/10.1016/j.otohns.2007.01.039
- [Background] Kallambettu V, Bae Y, Carrau R. Velopharyngeal Function Post Head and Neck Cancer: A Review. Ear Nose Throat J. 2024 Sep;103(9):NP567-NP577. doi: 10.1177/01455613211070895. Epub 2022 Jan 28. PMID 35081810
- [Background] Golding-Kushner KJ, Argamaso RV, Cotton RT, Grames LM, Henningsson G, Jones DL, Karnell MP, Klaiman PG, Lewin ML, Marsh JL, et al. Standardization for the reporting of nasopharyngoscopy and multiview videofluoroscopy: a report from an International Working Group. Cleft Palate J. 1990 Oct;27(4):337-47; discussion 347-8. doi: 10.1597/1545-1569(1990)0272.3.co;2. PMID 2253379
- [Background] Alfwaress F, Kummer AW, Weinrich B. Nasalance Scores for Normal Speakers of American English Obtained by the Nasometer II Using the MacKay-Kummer SNAP-R Test. Cleft Palate Craniofac J. 2022 Jun;59(6):765-773. doi: 10.1177/10556656211025406. Epub 2021 Jun 29. PMID 34184583